CLINICAL TRIAL: NCT04205500
Title: Treatment With Specific Carbohydrate Diet in Children With Juvenile Idiopathic Arthritis
Acronym: JIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other); Swedish University of Agricultural Sciences (Other)
Responsible Party: Principal Investigator, Lillemor Berntson, Associate professor, Uppsala University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2016/263
Record Dates: First submitted 2019-12-12; First posted 2019-12-19 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: juvenile; arthritis; diet
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with juvenile idiopathic arthritis (Experimental): The specific carbohydrate diet has been shown to have beneficial effects on IBD and has been implemented in Seattle Children's IBD centre, with some patients using SCD either as primary or complementary therapy. The SCD is a nutritionally balanced diet focused on removing many complex carbohydrates such as grains, dairy products except for yoghurt fermented over 24 hours, vegetables rich in starch and sugars except for monosaccharides like in honey. Participants can eat meat but since it has to be unprocessed food the investigator's experience is that the amounts of meat are not very big. Fish, eggs, sea-food is allowed. Bread is baked from nut and almond flour.
  Interventions: Other: Specific carbohydrate diet

INTERVENTIONS:
Other: Specific carbohydrate diet — Specific carbohydrate diet (see arm description)

SUMMARY:
The aim of this study is to explore if an already established diet with anti-inflammatory effect in paediatric inflammatory bowel disease would have an anti-inflammatory effect in children with JIA. The diet is called specific carbohydrate diet.

DETAILED DESCRIPTION:
Children classified with JIA, in a low-to-medium disease activity and without having changed DMARD or bDMARD in the last 12 weeks are included. Only motivated children and parents can participate. Before inclusion the family are informed orally about the study plan, the diet and practical issues regarding the study and they receive written information including for example a product list and a recipe booklet. A dietician and the principal investigator follows the child and parents during visits, by mail and phone. After the baseline visit, the family has two weeks to get used to the new diet. At baseline, after two, four and twelve weeks on the diet the child is examined, blood exams are performed and blood is stored at -70, fecal samples and urine is also collected. At inclusion and after four weeks saliva sample for bacteria is collected. The child fills in the child health assessment questionnaire, (CHAQ) for a score of the physical ability and DisabKids for an overall assessment of the childs well-being.

ELIGIBILITY:
Inclusion Criteria:

* Participants should fulfill criteria for JIA according to the ILAR criteria
* Participants should not be older than 16 years at onset of disease
* Participants should have a low-medium disease activity with an E-SR of 30 at the most and/or no more than two active joints at inclusion.
* DMARD and bDMARD should not have been changed within the last 12 weeks before inclusion.
* Any gastro- intestinal complaints should be investigated before inclusion.
* Fecal calprotectin should be normal.
* The child as well as the parents need to be motivated for the child to try a dietary intervention for at least four weeks, preferably longer.

Exclusion criteria:

* Children with the systemic category of JIA.
* Children with an unstable inflammatory situation with > 2 inflamed joints and/or an E-SR of more than 30.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in number of inflamed joints | At baseline compared to four weeks of intervention
  Physical examination
Change in CHAQ, child health assessment questionnaire | At baseline compared to four weeks of intervention
  A questionnaire for assessment of physical function, min-max, 0-3. A higher score means worse physical function
Change in overall well-being | At baseline compared to four weeks of intervention
  Global assessment visual analogue scale (VAS), for the patient min-max, 0-10 cm. A higher score means worse overall well-being
Change in assessment of pain: visual analogue scale | At baseline compared to four weeks of intervention
  Global assessment visual analogue scale (VAS) for Pain, min-max, 0-10 cm. A higher score means more pain
Change in assessment of morning stiffness | At baseline compared to four weeks of intervention
  Number of minutes

SECONDARY OUTCOMES:
Change in Microbiota in fecal samples | At baseline compared to four weeks of intervention
  16sSrRNA and Metagenomics
Change in Short chain fatty acids in fecal samples | At baseline compared to four weeks of intervention
  Analysed, using a HPLC-machine, Agilent technology 1100-series, presented in mg/gr

CONTACTS AND LOCATIONS:
Overall Officials: Lillemor Berntson, Ass Prof, Principal Investigator — Unit of Pediatric Rheumatology, Akademiska hospital, Uppsala University, Sweden
Locations (1):
- Unit of Pediatric Rheumatology, Akademiska hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Berntson L. A pilot study of possible anti-inflammatory effects of the specific carbohydrate diet in children with juvenile idiopathic arthritis. Pediatr Rheumatol Online J. 2021 Jun 10;19(1):88. doi: 10.1186/s12969-021-00577-3. PMID 34112181